CLINICAL TRIAL: NCT02971384
Title: Controlled, Randomized, Double-blind, Multicentre Study on Efficacy and Safety of Echinaforce Junior Tablets in Comparison With Vitamin C for the Prevention of Viral Respiratory Tract Infections in Children (4-12 Years)
Brief Title: Echinacea Junior vs Vitamin C in Children 4-12 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A. Vogel AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 5000120
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2017-12

CONDITIONS: Respiratory Tract Infection Viral
MeSH Terms: interventions — Echinaforce; Echinacea extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Echinaforce Junior Tablets (Experimental): Hydroalcoholic extract of Echinacea purpurea herb and radix
  Interventions: Drug: Echinaforce
- Vitamin C Tablets (Active Comparator): synthetically produced ascorbic acid
  Interventions: Drug: Echinaforce

INTERVENTIONS:
Drug: Echinaforce
  Other Names: Echinacea purpurea

SUMMARY:
Aim of this study is to investigate efficacy and safety of Echinaforce Junior Tablets (250mg) in comparison with Vitamin C tablets in the prevention of acute viral respiratory tract infections.

DETAILED DESCRIPTION:
200 children aged 4-12 years are recruited by pediatricians and general practitioners and are allocated to preventive treatment with either Echinaforce Junior tablets or Vitamin C. Children take 3 x 1 tablet per day over a period of 2 months followed by 1 week treatment break and an intermediate study visit (V2). Thereafter children continue with preventive Treatment for another 2 months, followed by exclusion visit (V3).

Parents are required to contact a study coordinator at the occurrence of acute respiratory Symptoms to initiate symptom recording via internet-based e-diary. On day 1 - 3 of episode parents will sample nasal secretion, which will be analysed for common respiratory agents.

ELIGIBILITY:
Inclusion Criteria:

* 4-12 years
* written informed consent by parents and optionally by child
* daily Access to computer/email
* german language skills

Exclusion Criteria:

* 13 years or older, younger than 4 years
* participation in a clinical study during past 30 days
* intake of antimicrobial, antiviral, immunosuppressive substances, salicylic medicaments (like Aspirin)
* surgical intervention 3 months Prior to inclusion or planned intervention during the observation period
* known Diabetes mellitus
* known and treated atopy or Asthma
* cystic fibrosis, bronchopulmonary dysplasia, chronic obstructive pulmonary disease (COPD)
* diseases of the immunosystem (like autoimmune disorders, degenerative illnesses (like AIDS or leucosis))
* Metabolic or Resorption disorders
* Liver or kidney diseases
* Serious health Problems (e.g. neurological Problems)
* known allergies against compositae (e.g. camomile or dandelion) or any of the substances of the investigational product

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
cumulative number of cold days | 4 months prevention
  total number of days with cold symptoms as per diary entries

SECONDARY OUTCOMES:
Occurrence of adverse events | 4 months prevention
  Occurrence of adverse events will be analysed by descriptive methods
Analysis of duration and severity of respiratory episodes (single Symptoms and total symptom score) | 4 months prevention
  Patients will rate respiratory symptoms in a diary at occurrence of acute respiratory tract infections and the entries will be analysed descriptively for the two treatment groups
Incidence of respiratory tract infections (viral RTIs) | 4 months prevention
  Occurrence of colds and flu episodes
Acceptance in the view of the parents | 4 months prevention
  Parents will judge the acceptance after 4 months (would you use the medicament again?)
Occurrence of adverse drug reactions | 4 months prevention
  Occurrence of adverse drug reactions will be analysed by descriptive methods
Tolerability in view of the physician | 4 months prevention
  physicians will judge tolerability as "bad", "moderate", "good" or "very good"
Tolerability in view of the parents | After 4 months prevention
  parents will judge the tolerability after 2 and 4 months treatment as "bad", "moderate", "good" or "very good"
Efficacy in the view of the parents/children | 4 months prevention
  Parents/children will give their subjective impression of efficacy by ratings "bad", "moderate", "good" or " very good".
accompanying virus analytics | 4 months prevention
  nasal samples will be taken at occurrence of cold Symptoms and will be analysed for the presence of respiratory viruses
effects on the endogenous defense | 4 months prevention
  Question will be asked " do you think that the prevention had the follwing effects on the endogenous defense in your child?" (unchanged; improved; significantly improved")
Concomitant treatment and therapies | 4 months prevention
  Concomitant treatment and therapies will be coded using medical dictionary for Regulatory Agencies and will be analysed descriptively for the two treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Ogal, Dr. med., Principal Investigator — Arztpraxis für Kinder und Jugendliche
Locations (1):
- Dr. med. Mercedes Ogal, Brunnen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ogal M, Johnston SL, Klein P, Schoop R. Echinacea reduces antibiotic usage in children through respiratory tract infection prevention: a randomized, blinded, controlled clinical trial. Eur J Med Res. 2021 Apr 8;26(1):33. doi: 10.1186/s40001-021-00499-6. PMID 33832544